CLINICAL TRIAL: NCT05777512
Title: A Randomized Controlled Crossover Trial of Postpyloric Versus Gastric Feedings to Improve Pulmonary Outcomes in High-risk Preterm Infants
Brief Title: Randomized Controlled Crossover Trial of Postpyloric Feedings to Improve Pulmonary Outcomes in High-risk Preterm Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Jonathan Levin, Instructor of Pediatrics, Boston Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-P00043302
Record Dates: First submitted 2023-02-09; First posted 2023-03-21 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Chronic Lung Disease of Prematurity; Postpyloric Feeding; Nasojejunal Feeding; Bronchopulmonary Dysplasia; GERD; Gastro-esophageal Reflux
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: This is a randomized single crossover study design, with each of two 10-day study blocks. Infants will be individually randomized to the study intervention (jejunal feeding) in Block 1 or Block 2. The first 48 hours of each study block will be considered run-in/washout periods.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Gastric Followed by Jejunal Feeds (Experimental): Participants randomized into this group will begin with one ten-day block of nasogastric (NG) feeds followed by one ten-day block of nasojejunal (NJ, postpyloric) feeds.
  Interventions: Procedure: Gastric Feeds; Procedure: Jejunal Feeds
- Group B: Jejunal Followed by Gastric Feeds (Experimental): Participants randomized into this group will begin with one ten-day block of nasojejunal (NJ, postpyloric) feeds followed by one ten-day block of nasogastric (NG) feeds.
  Interventions: Procedure: Gastric Feeds; Procedure: Jejunal Feeds

INTERVENTIONS:
Procedure: Gastric Feeds — The participant will receive nutrition via a nasogastric tube. Gastric feedings will be administered as bolus feeds every 3 hours over 1 hour. Infants who are deemed able to advance oral feedings via mouth during the study period will be permitted to do so, and this will be recorded.
  Other Names: Nasogastric Feeding; NG feeds
Procedure: Jejunal Feeds — The participant will receive nutrition via a nasojejunal tube. Postpyloric feedings will be administered continuously into the jejunum. Infants who are deemed able to advance oral feedings via mouth during the study period will be permitted to do so, and this will be recorded.
  Other Names: Nasojejunal Feeding; Postpyloric Feeding; NJ Feeds

SUMMARY:
The purpose of this study is to determine if postpyloric feedings effectively improve objective measures of pulmonary health in preterm infants with chronic lung disease when compared with nasogastric (NG) feedings. This research will (1) determine the optimal nutritional management to prevent a common and costly complication of prematurity, and (2) use a novel crossover design that examines outcomes of clinical endpoints alongside biomarkers.

DETAILED DESCRIPTION:
Bronchopulmonary dysplasia (BPD) affects up to 50,000 preterm infants annually in the United States and is the most common complication of prematurity. Despite improving survival in preterm infants, incidence of BPD is increasing. Overall, 11% of infants are born preterm in the United States annually. While many outcomes of prematurity, including survival, have improved over time, the incidence of BPD has increased.

Nearly all babies with BPD require provision of feeds via an enteral tube due to feeding immaturity and ongoing need for respiratory support, and up to ¼ of babies with the most severe forms of BPD require this long-term, and are discharged home with nasal or surgically placed feeding tubes. However, enteral feeding into the stomach frequently results in reflux in preterm infants. This may cause aspiration into the respiratory tract, which can result in further damage to the lungs and worsen respiratory outcomes.

The study will measure the impact of NJ feedings on lung disease severity in a prospective crossover trial among infants at high-risk of developing BPD.

Each randomized patient will participate in two blocks of feeding, a nasogastric (NG) and a nasojejunal (NJ, postpyloric) block. Subjects will be randomized to either the control (NG) or intervention (NJ) feedings in the first block. Outcomes will be compared pairwise by subject between the NG and NJ blocks.

The findings of this study would be immediately impactful for neonatologists, pediatricians, pediatric pulmonologists, pediatric gastroenterologists, advanced practitioners, and nutritionists who determine nutritional strategies for preterm infants.

ELIGIBILITY:
Inclusion Criteria:

Preterm infants born < 32 weeks' gestation may enroll at 34-44 weeks post-menstrual age, who:

1. Remain on either invasive ventilation or non-invasive ventilation (continuous positive airway pressure or nasal intermittent positive pressure ventilation) for minimum 48 hours at the time of study entry. The minimum support required for inclusion is CPAP > 5cm H2O or CPAP 5 with FiO2 > 21%.
2. Have ongoing need for respiratory support due to underlying lung disease from prematurity.
3. Are tolerating > 80 ml/kg/day of enteral feedings at baseline, either via nasogastric (NG) or nasojejunal (NJ) tube. Patients may be receiving gastric (NG) or postpyloric (NJ) feedings.

Exclusion Criteria:

1. Infants who are transiently on respiratory support at the time of study entry due to another reason than underlying lung disease from prematurity; for example, recovery from a surgical intervention.
2. Infants who have other comorbidities that significantly contribute to lung disease, including cyanotic congenital heart disease, or other genetic, congenital, or pulmonary abnormalities.
3. Infants who were evaluated for necrotizing enterocolitis (including holding feedings) in the 7 days prior to study enrollment.
4. Infants with known gastrointestinal or airway malformations that would affect tolerance of feeds or the route of delivery of enteral feedings.

Ages: 0 Hours to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in modified respiratory severity score (mRSS) | Over a 15 day period during study participation
  mRSS is a validated measurement for respiratory severity in chronic lung disease in neonates.
Tracheal Aspirates | Over a 15 day period during study participation.
  For infants who remain on invasive respiratory support, the study team will collect tracheal aspirates for the measurement of bile acid and pepsin concentration.

SECONDARY OUTCOMES:
Respiratory Support Over the Course of the Study | Over a 15 day period during study participation
  The study team will monitor the patient's respiratory support needs by reviewing the medical record.
Nutritional Status Over the Course of the Study | Over a 15 day period during study participation
  The study team will monitor the patient's nutritional status by reviewing the medical record at the end of each study period.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Levin, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No